CLINICAL TRIAL: NCT03314324
Title: A Study of Patient Preference Between ODM-201 and Enzalutamide in Men With Metastatic Castrate-resistant Prostate Cancer
Acronym: ODENZA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2017-001606-14; 2017/2555 (Other: CSET number)
Record Dates: First submitted 2017-10-13; First posted 2017-10-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castrate-resistant Prostate (CRPC) Cancer
MeSH Terms: conditions — Neoplasms | interventions — darolutamide; enzalutamide

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label, multicenter, cross-over phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ODM-201 (Experimental)
  Interventions: Drug: ODM-201
- Enzalutamide (Active Comparator)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: ODM-201 — ODM-201: 600 mg (2 x 300 mg tablets) twice daily with food equivalent to a total daily dose of 1200 mg. ODM-201 should be taken at similar times day, approximately 12 hours between doses.
  Arms: ODM-201
Drug: Enzalutamide — Enzalutamide: 160 mg/day (4 x 40 mg tablets) taken once a day preferably with food, preferably in the evening (Enzalutamide can generally be given with or without food, but in the present trial, it is preferable that it is given with food, to be consistent with ODM-201 intake).
  Arms: Enzalutamide

SUMMARY:
To assess patient preference between ODM-201 and enzalutamide by patient preference questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Male patients older than 18 years
* Histologically confirmed adenocarcinoma of the prostate
* Evidence of metastatic disease (imaging can include bon scan, CT scan, PET choline, PET PSMA and MRI)
* Continued androgen deprivation therapy (ADT) either with LHRH agonists/antagonists or bilateral orchiectomy
* Serum testosterone <0.50 ng/ml (1.7 nmol/L)
* Progressive disease (PSA progression or radiological progression or clinical progression) as per PCWG3 criteria
* ECOG 0-1 (2 is accepted if the impairment is not due to prostate cancer)
* Asymptomatic or mildly symptomatic prostate cancer as measured on the Brief Pain Inventory Short Form question 3 (i.e. worst pain in the last 24 hours <4 on a Visual Analog Scale)
* Information imparted to the patient and the informed consent form signed by the patient or his legal representative
* Ability to comply with the protocol procedures
* Patient affiliated to a social security system or beneficiary of the same
* Sexually active male subjects unless surgically sterile, must agree to use condoms as an effective barrier method and refrain from sperm donation, and/or their female partners of reproductive potential to use a method of effective birth control, during the study treatment and for 3 months after the end of the treatment
* adequate organ or bone marrow function as evidenced by:
* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count ≥ 1.5 x 109/L,
* Platelet count ≥ 100 x 109/L, (subject must not have received any growth factor within 4 weeks or blood transfusion within 7 days of the hematology laboratory sample obtained at screening)
* AST/SGOT and/or ALT/SGPT ≤1.5 x ULN;
* Total bilirubin ≤ 1.5 x ULN, (except subjects with a diagnosis of Gilbert's disease),
* Serum creatinine ≤ 2 x ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to the CKDEPI formula and patients with creatinine clearance <60 mL/min should be excluded.

Exclusion Criteria:

* Prior treatment with abiraterone, enzalutamide, ODM-201, ARN- 509 or any other next-generation AR axis-targeting drug
* Prior treatment with a taxane for CRPC (prior treatment with a taxane for castration-sensitive or castration-naïve prostate cancer is allowed)
* Prior treatment with radium-223
* Patients receiving an investigational drug within 4 weeks prior to enrolment (approved drugs with a long history of use such as aspirin, statins, heparins, or metformin, even used in an experimental setting are accepted)
* Treatment with radiotherapy (external beam radiation therapy [EBRT], brachytherapy, or radiopharmaceuticals) within 2 weeks before randomization
* Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs
* Acute toxicities of prior treatments and procedures not resolved to grade <=1 or baseline before randomisation.
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure (New York Heart Association (NYHA) Class III or IV)
* Uncontrolled hypertension as indicated by a resting systolic blood pressure (BP) ≥160 mmHg or diastolic BP ≥100 mmHg despite optimal medical management
* Had a prior malignancy. Adequately treated basal cell or squamous cell carcinoma of skin or superficial bladder cancer that has not spread behind the connective tissue layer (i.e., pTis, pTa, and pT1) is allowed, as well as any other cancer for which treatment has been completed ≥5 years before randomization and from which the subject has been disease-free
* A gastrointestinal disorder or procedure which is expected to interfere significantly with absorption of study treatment
* An active viral hepatitis, active human immunodeficiency infection(HIV), or chronic liver disease with a need for treatment.
* Any other serious or unstable illness or infection, or medical, social, or psychological condition, that could jeopardize the safety of the subject and/or his compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results
* Inability to swallow oral medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Patient preference | up to 24 months
  Patient preference (assessed by a single question) between ODM-201 and enzalutamide after completion of the second period of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided